CLINICAL TRIAL: NCT04157777
Title: THE EFFECT OF PERİNEUM MASSAGE WİTH OLİVE OİL
Brief Title: THE EFFECT OF PERİNEUM MASSAGE WİTH OLİVE OİL ON PERİNEUM INTEGRİTY AND DURATİON OF SECOND PERİOD OF DELİVERY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Evrim Bayraktar, Assoc Prof., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Erciyes U
Record Dates: First submitted 2019-10-15; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Prevention
Keywords: Perineum massage, perineal trauma,perineal laceration
MeSH Terms: interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- massage (Experimental): Among women who applied to Maternity Hospital 350 pregnant women were assigned to massage group. Participants in massage group filled out an information form including socio-demographic characteristics. Perineum massage with olive oil in the second period of delivery was performed to massage group.In massage group when they progressed to full dilatation of the cervix, the midwife inserted two fingers inside vagina and using a sweeping motion gently stretched the perineum with lubricant 5 up to 10 minutes, in and between mother's pushing in the second stage of labour.
  Interventions: Other: Perineum massage with olive oil
- control (Experimental): Among women who applied to Maternity Hospital 350 pregnant women were assigned to control group. Participants in control group filled out an information form including socio-demographic characteristics.And, no other interventions except for applications performed routinely in the delivery room were done.In control group just Ritgen Maneuver was applied. At last, we com-pared the rate of intact perineum, episiotomy and laceration, mean duration of the second stage of labor and Apgar score in 1 and 5 minutes be-tween two groups.
  Interventions: Other: Perineum massage with olive oil

INTERVENTIONS:
Other: Perineum massage with olive oil — Descriptive form used for data collection included questions about women's sociodemographic features, medical and obstetric history and previous and present birthsof women participated in the study.
  The Reeda Scale The scale is consisted of five parameters of healing: Redness, Edema, Ecchymosis, Discharge Approximation.
  Pregnant women who came to the delivery room and met the criteria were randomly selected and assigned to experimental and control group according to age and educational status.
  There was not any change in the birth process of the delivery room during data collection and the pregnant women received routine care and treatments.
  REEDA scale was administered by other midwives who worked at the puerperal room where pregnant women stayed after birth and did not know their groups because those who gave vaginal birth were early discharged from the hospital as they could answer only the first three parameters of REEDA scale.

SUMMARY:
Aims and objectives:This experimental study was conducted to determine the effect of perineum massage with olive oil performed in the second period of the delivery on travay duration, episiotomy requirement and perineum tears in term pregnant women.

Background: Perineal trauma that may occur during labor may pose a critical risk both for mother's health and her quality of life.

Design: A randomized controlled trial. This study adhered to CONSORT 2010 checklist guidelines for qualitative research reporting Method: Among women who applied to Maternity Hospital 350 pregnant women were assigned to massage group while other 350 were to control group. Participants in both groups filled out an information form including socio-demographic characteristics. Perineum massage with olive oil in the second period of delivery was performed to massage group. In the control group, no other interventions except for applications performed routinely in the delivery room were done.

Results: Episiotomy was done in 34.3% of massage group while in 48.6% of control group. Percentage of being performed episiotomy in the massage group significantly decreased (p<0.05).Tear appeared in 17.7% of the massage group while in 38.0% of the controls. Percentage of tear formation in the massage group significantly decreased (p<0.05). No statistically significant difference was found between the second period of the delivery of massage and control group. All of the pregnant women in the massage group and midwives who performed massage were satisfied with perineum massage with olive oil in the delivery and stated that they would suggest and perform this application Conclision: Regarding the results of this study and those of other studies, perineal massage during the second stage of labor can reduce the need for episiotomy, and avoid perineal injuries, and perineal pain.

This study provides useful information to clinician and researchers when determining practices such as postnatal standing up in early period,reduced episiotomy requirement, mother's health ,her quality of life, shorter hospital stay and perineal trauma.

What does this paper contribute to the wider global clinical community?

* Perineum massage performed with olive oil in delivery are an effective, inexpensive, simple, and well-tolerated way to improve intact perineum..
* Perineum massage performed with olive oil in delivery are safe and associated with mother's health and her quality of life and shorter hospital stay.

DETAILED DESCRIPTION:
The idea that birth process should be undergone minimal intervention has been spreading. Unlike the abovementioned idea, the fact that episiotomy practice -especially on the primiparous pregnant women- has almost been a routine in Turkey and it has been practiced -even if it is not necessary- despite the fact that itprolongs the post-partum healing and increases perineum trauma risks.

Perineal trauma is described as the damage that occurs spontaneously or due to a surgical incision or episiotomy during the labor in the genital region. Perineal trauma that may occur during labor may pose a critical risk both for mother's health and her quality of life. Perineal trauma is accompanied with short term or long term morbidity during and after birth and affects sexuality and physical image of the women negatively. Some of these effects are painful sexual intercourse, fecal and urinary incontinence and continuous perineal pain.

Perineal massage performed by using an oily substance that has lubricant properties is described as the massage made on the muscles around the vagina and its tissues. The massage,which is thought to haveimportant effects onelasticity of the tissues and muscles and the rehabilitation is thought to provide benefits for vaginal births due to the similar useful effects on the tissues and muscles around the perineal. Perineal massage with lubricant is a poten-tial therapeutic approach implemented at the second stage of delivery.

Background Perineal tissues should be pulled aside to allow the neonate exit from the vagina.Studies regarding the perineal pulling and massaging in the second stage of labor for relaxing the perineum and possibly preventing perineal laceration and episiotomy, have concluded that the perineal pulling and massaging increase possibility of childbirth with an intact perineum. Perineal massage increases elasticity and blood supply to the perineum and leads to easier pulling and less pain during childbirth. It also reduces the possibility of perineal laceration, the need to episiotomy, and postpartum perineal pain.

Aims:

The aim of the present research was to determine the effects of massage performed by using olive oil on travail duration, episiotomy requirement and perineal tears for the term pregnancies during second stage of the labor.

COLLOUT: Perineal trauma that may occur during labor may pose a critical risk both for mother's health and her quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women who had cephalic presentation
* with vertex presentation
* alive primiparous pregnancy at 38-40thgestational weeks (according to last menstruation date or ultrasonography determination)
* They also did not have any cesarean or any kind of uterine surgical operation
* aged between 17 and 40
* with no risk factors (heart disease, placenta praevia, oligohydramnios, preeclampsia, anhydramnios, diabetes, epilepsy), multiparous≤ three times, literate and without counter indication for vaginal birth were included in the research.

Exclusion Criteria:

* history of any cesarean operation or uterus surgery
* dead fetus, vaginal bleeding with no explanation
* twin pregnancy
* presence of fetal anomaly
* estimated fetal weight over 4500 gr. as determined by ultrasonography and presence of presentation anomaly.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2009-03-15 (Actual); Primary Completion 2010-04-09 (Actual); Study Completion 2011-04-16 (Actual)

PRIMARY OUTCOMES:
episiotomy requirement and perineal tears for the term pregnancies | The midwives were told to perform the massage after the pregnant woman was placed in the obstetric table and her cervical dilatation was between 7 and 10 cm.
  Perineal massage performed byusing an oily substance that has lubricant properties is described as the massage made on the muscles around the vagina and its tissues. The massage,which is thought to haveimportant effects onelasticity of the tissues and muscles and the rehabilitation is thought to provide benefits for vaginal births due to the similar useful effects on the tissues and muscles around the perineal3-6.The aim of the present research was to determine the effects of massage performed by using olive oil on travail duration, episiotomy requirement and perineal tears for the term pregnancies .

SECONDARY OUTCOMES:
during second stage of the labor. | The midwives were told to perform the massage after the pregnant woman was placed in the obstetric table and her cervical dilatation was between 7 and 10 cm.
  Perineal massage performed byusing an oily substance that has lubricant properties is described as the massage made on the muscles around the vagina and its tissues. The massage,which is thought to haveimportant effects onelasticity of the tissues and muscles and the rehabilitation is thought to provide benefits for vaginal births due to the similar useful effects on the tissues and muscles around the perineal.The aim of the present research was to determine the effects of massage performed by using olive oil on travail duration, episiotomy requirement and perineal tears for the term pregnancies during second stage of the labor.

IPD SHARING:
Plan to Share IPD: No